CLINICAL TRIAL: NCT06691113
Title: A Randomized, Double-blind, Placebo-controlled, Proof-of-Concept (PoC) Study to Assess the Efficacy, Safety and Tolerability of Itepekimab in Participants With Inadequately Controlled Chronic Rhinosinusitis Without Nasal Polyps
Brief Title: A Proof-of-Concept Study to Assess the Efficacy, Safety and Tolerability of Itepekimab (Anti--IL-33 mAb) in Participants With Chronic Rhinosinusitis Without Nasal Polyps
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT18421; 2024-515576-12 (Registry Identifier: CTIS); U1111-1306-6643 (Registry Identifier: ICTRP)
Record Dates: First submitted 2024-11-12; First posted 2024-11-15 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Chronic Rhinosinusitis Without Nasal Polyps
MeSH Terms: interventions — itepekimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Itepekimab high dose (Experimental): Subcutaneous (SC) administration of Itepekimab high dose for 24 weeks
  Interventions: Drug: Itepekimab (SAR440340); Drug: Mometasone furoate nasal spray (MFNS)
- Itepekimab low dose (Experimental): SC administration of Itepekimab low dose for 24 weeks
  Interventions: Drug: Itepekimab (SAR440340); Drug: Placebo; Drug: Mometasone furoate nasal spray (MFNS)
- Placebo (Placebo Comparator): SC administration of matching placebo for 24 weeks
  Interventions: Drug: Placebo; Drug: Mometasone furoate nasal spray (MFNS)

INTERVENTIONS:
Drug: Itepekimab (SAR440340) — Pharmaceutical form: Solution for injection in prefilled syringe. Route of administration: Subcutaneous
  Other Names: REGN3500
  Arms: Itepekimab high dose; Itepekimab low dose
Drug: Placebo — Pharmaceutical form: Solution for injection in prefilled syringe. Route of administration: Subcutaneous
  Arms: Itepekimab low dose; Placebo
Drug: Mometasone furoate nasal spray (MFNS) — Pharmaceutical form: Solution for administration via spray pump. Route of administration: Intranasal spray

SUMMARY:
ACT18421 is a multinational, randomized, double-blind, placebo-controlled, parallel-group, Phase 2 study with 3 treatment groups. The purpose of the study is to evaluate the efficacy, safety and tolerability of 2 dosing regimens of itepekimab compared to placebo in male and female participants with chronic rhinosinusitis without nasal polyps (CRSsNP) aged 18 years of age and older.

Study details include:

* The study duration (4-week screening, 24--week intervention, 20--week safety followup) will be 48 weeks.
* The intervention duration will be 24 weeks.
* The number of visits will be 7 site visits and 8 phone/remote visits.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 years of age or older.
* Participants must have ongoing symptoms of nasal congestion/obstruction at least 12 consecutive weeks before Visit 1 and a Nasal Congestion Score (NCS) ≥2 at Visit 1 (day score) and Visit 2 (weekly average score).
* Participants must have sinus Total Symptom Score (sTSS) (NC, rhinorrhea, facial pain/pressure) ≥5 at Visit 1 (day score) and Visit 2 (weekly average score).
* Participants must have at least one of the following features:

  * Prior sinonasal surgery (as protocol defined) for chronic rhinosinusitis (CRS).
  * Treatment with systemic corticosteroid(s) (SCS) within the prior 2 years before Screening (Visit 1)
  * Worsening symptoms of CRS in the past 2 years which would have required treatment with SCS, however participant is intolerant or has a contraindication to SCS.
* Participants must have bilateral inflammation of paranasal sinuses with bilateral ethmoid and maxillary opacification on screening CT scan. Participants must have ≥25% opacification of the ethmoid sinuses and ≥25% opacification of at least 1 maxillary sinus by central reading of CT scan.
* Participants must have a Sino-Nasal Outcome Test-22-Items (SNOT-22) score of ≥20 at Visit 1 and Visit 2.
* Participants who have received a stable dose of mometasone furoate nasal spray (MFNS) for at least 3 weeks before Visit 2.
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least 1 of the following conditions applies:

  * Is not a women of childbearing potential (WOCBP). OR
  * Is a WOCBP and agrees to use a contraceptive method that is highly effective, with a failure rate of <1% during the study (at a minimum until 20 weeks after the last dose of study intervention).

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Participants with conditions/concomitant diseases making them non-evaluable at Visit 1 or for the primary efficacy endpoint.
* Participants with nasal cavity malignant tumor and benign tumors (eg, papilloma, blood boil).
* Radiological suspicion or confirmed invasive or expansive fungal rhinosinusitis.
* Have any clinically significant diseases or disorders (eg, cardiovascular, pulmonary, gastrointestinal, liver, kidney, neurological, musculoskeletal, endocrine, metabolic, psychiatric, physical impairment) that, in the opinion of the Investigator, may put the subject at risk by participating in the study, or interfere with the subject's intervention, assessment, or influence the results of the study, or have compliance issues with the study.
* Sinus surgery within 6 months before Screening (Visit 1)
* Participants who received SCS 1 month prior to Screening (Visit 1) or during the screening period (between Visit 1 and Visit 2).
* Participants treated with other intranasal corticosteroid(s) (INCS) (only study provided AxMP [MFNS] is permitted), intranasal emitting devices/stents, nasal spray using exhalation delivery system such as Xhance™ during the screening period.
* Participants with a history of severe systemic hypersensitivity reaction to mAb.
* Known allergy to itepekimab or to its excipients. Any drug or other allergy that, in the opinion of the Investigator, contraindicates participation in the study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2026-08-07 (Estimated); Study Completion 2027-02-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in sinus (maxillary, ethmoid) percent opacification volume assessed by CT scan | Baseline to End of Treatment (EOT) (Week 24)
  Change from baseline in sinus inflammation as assessed by Computerized Tomography (CT) scan of the sinuses in the itepekimab-- compared to placebo-- treated study participants on the background of intranasal corticosteroid (INCS).

SECONDARY OUTCOMES:
Change from baseline in the sTSS | Baseline to EOT (Week 24)
  The CRSsNP sinus Total Symptom Score (sTSS) is a composite score derived from nasal congestion (NC), anterior/posterior rhinorrhea, and facial pain/pressure. The total score ranges from 0 to 9 with higher scores indicating greater overall symptom severity.
Change from baseline in nasal congestion (NC) severity score using the CRSsNP daily ediary | Baseline to EOT (Week 24)
  The CRSsNP sinonasal symptom diary is designed to assess the severity of CRS sinonasal symptoms on daily basis. These symptoms include NC/obstruction, anterior rhinorrhea and posterior rhinorrhea, facial pain/pressure, loss of smell, and headache. Each of the individual items of the diary are scored from 0 ("No symptoms") to 3 ("Severe symptoms - symptoms that are hard to tolerate, cause interference with activities or daily living"). Higher scores on the items of the individual symptoms denote greater symptom severity.
Change from baseline in anterior/posterior rhinorrhea severity score using the CRSsNP daily ediary | Baseline to EOT (Week 24)
  The CRSsNP sinonasal symptom diary is designed to assess the severity of CRS sinonasal symptoms on daily basis. These symptoms include NC/obstruction, anterior rhinorrhea and posterior rhinorrhea, facial pain/pressure, loss of smell, and headache. Each of the individual items of the diary are scored from 0 ("No symptoms") to 3 ("Severe symptoms - symptoms that are hard to tolerate, cause interference with activities or daily living"). Higher scores on the items of the individual symptoms denote greater symptom severity.
Change from baseline in facial pain/pressure severity score using the CRSsNP daily ediary | Baseline to EOT (Week 24)
  The CRSsNP sinonasal symptom diary is designed to assess the severity of CRS sinonasal symptoms on daily basis. These symptoms include NC/obstruction, anterior rhinorrhea and posterior rhinorrhea, facial pain/pressure, loss of smell, and headache. Each of the individual items of the diary are scored from 0 ("No symptoms") to 3 ("Severe symptoms - symptoms that are hard to tolerate, cause interference with activities or daily living"). Higher scores on the items of the individual symptoms denote greater symptom severity.
Change from baseline in loss of smell severity score using the CRSsNP daily ediary | Baseline to EOT (Week 24)
  The CRSsNP sinonasal symptom diary is designed to assess the severity of CRS sinonasal symptoms on daily basis. These symptoms include NC/obstruction, anterior rhinorrhea and posterior rhinorrhea, facial pain/pressure, loss of smell, and headache. Each of the individual items of the diary are scored from 0 ("No symptoms") to 3 ("Severe symptoms - symptoms that are hard to tolerate, cause interference with activities or daily living"). Higher scores on the items of the individual symptoms denote greater symptom severity.
Change from baseline in SNOT-22 total score | Baseline to EOT (Week 24)
  The Sino-Nasal Outcome Test-22-Items (SNOT-22) is a patient-reported outcome questionnaire designed to assess the impact of chronic rhinosinusitis (CRS) on patients' Health-Related Quality of Life (HRQoL). It has 22 items covering symptoms, social/emotional impact, productivity, and sleep consequences of CRS. A global score ranges from 0 to 110 with higher score indicating greater rhinosinusitis-related health burden.
Change from baseline in sinus opacification as measured by the Lund-Mackay (LMK) score and the modified LMK score | Baseline to EOT (Week 24)
  The LMK and the modified LMK scoring systems are based on points given for degree of opacification, which are applied to the maxillary, anterior ethmoid, posterior ethmoid, sphenoid, frontal sinus on each side. The osteomeatal complex is graded as 0 = not occluded, or 2 = occluded, deriving a maximum score of 12 per side.
Incidence of treatment-emergent adverse events (TEAEs), treatment-emergent adverse events of special interest (TEAESIs), treatment emergent serious adverse events (TESAEs), and TEAEs leading to intervention discontinuation | Baseline up to End of Study (EOS) (Week 44)
Itepekimab concentration in serum | Baseline to EOS (Week 44)
Incidence of treatment-emergent (TE) anti-itepekimab antibodies responses | Baseline to EOS (Week 44)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (57):
- United States (10):
  - Allervie Clinical Research - Birmingham- Site Number : 8400006, Birmingham, Alabama
  - Modena Allergy + Asthma- Site Number : 8400005, La Jolla, California
  - United Medical Doctors - Murrieta- Site Number : 8400001, Murrieta, California
  - Sacramento Ear Nose & Throat - Roseville- Site Number : 8400008, Roseville, California
  - Western States Clinical Research- Site Number : 8400009, Wheat Ridge, Colorado
  - Advanced Research Associates (ARA) Professionals- Site Number : 8400002, Miami, Florida
  - Treasure Valley Medical Research- Site Number : 8400022, Boise, Idaho
  - ENT Associates of Texas - McKinne- Site Number : 8400013, McKinney, Texas
  - Alamo ENT Associates- Site Number : 8400026, San Antonio, Texas
  - Eastern Virginia Medical School (EVMS) Medical Group- Site Number : 8400007, Norfolk, Virginia
- Argentina (3):
  - Investigational Site Number : 0320003, San Miguel de Tucumán, Tucumán Province
  - Investigational Site Number : 0320001, Buenos Aires
  - Investigational Site Number : 0320004, Corrientes
- Belgium (4):
  - Investigational Site Number : 0560003, Brussels
  - Investigational Site Number : 0560004, Gesves
  - Investigational Site Number : 0560002, Ghent
  - Investigational Site Number : 0560001, Leuven
- Canada (6):
  - Investigational Site Number : 1240005, London, Ontario
  - Investigational Site Number : 1240002, Montreal, Quebec
  - Investigational Site Number : 1240001, Québec, Quebec
  - Investigational Site Number : 1240003, Québec, Quebec
  - Investigational Site Number : 1240012, Québec, Quebec
  - Investigational Site Number : 1240009, Trois-Rivières, Quebec
- Chile (3):
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Concepción, Región del Biobío
- China (4):
  - Investigational Site Number : 1560004, Baotou
  - Investigational Site Number : 1560001, Beijing
  - Investigational Site Number : 1560002, Shanghai
  - Investigational Site Number : 1560003, Zibo
- France (4):
  - Investigational Site Number : 2500012, La Rochelle
  - Investigational Site Number : 2500004, Marseille
  - Investigational Site Number : 2500005, Montpellier
  - Investigational Site Number : 2500010, Poitiers
- Italy (3):
  - Fondazione Policlinico Universitario Campus Bio-Medico-Site Number : 3800002, Rome, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Site Number : 3800001, Rome, Roma
  - Azienda Ospedaliero-Universitaria Pisana-Site Number : 3800003, Pisa
- Poland (5):
  - Investigational Site Number : 6160002, Poznan, Greater Poland Voivodeship
  - Investigational Site Number : 6160006, Krakow, Lesser Poland Voivodeship
  - Investigational Site Number : 6160008, Lodz, Lódzkie
  - Investigational Site Number : 6160001, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160004, Bielsko-Biala, Silesian Voivodeship
- Portugal (2):
  - Investigational Site Number : 6200001, Guimarães
  - Investigational Site Number : 6200002, Porto
- Romania (2):
  - Investigational Site Number : 6420001, Brasov
  - Investigational Site Number : 6420002, Bucharest
- South Korea (5):
  - Investigational Site Number : 4100005, Cheonan-si, Chungcheongnam-do
  - Investigational Site Number : 4100003, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100004, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
- Spain (6):
  - Investigational Site Number : 7240003, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240002, L'Hospitalet de Llobregat, Catalunya [Cataluña]
  - Investigational Site Number : 7240004, Jerez de la Frontera, Cádiz
  - Investigational Site Number : 7240005, Pamplona, Navarre
  - Investigational Site Number : 7240001, Seville, Sevilla
  - Investigational Site Number : 7240006, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: ACT18421 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26272&tenant=MT_SNY_9011